CLINICAL TRIAL: NCT03574870
Title: Feasibility Study of a Wearable Sensor for Acquisition of Biometric Data in Head and Neck Cancer Patients During Locoregional Therapy
Brief Title: Wearable Sensor for Biometrics During Locoregional Therapy for Head and Neck Cancer
Acronym: FITBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU 102016-059
Record Dates: First submitted 2018-05-18; First posted 2018-07-02 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Chemoraditherapy (Experimental): Patients with head and neck cancer require chemo and radiation therapy (Cohort A):
  A wearable sensor device will be issued at the time of trial enrollment. Patients will be instructed to wear the device on their wrist for 23 hours per day, 7 days per week, from the time of their radiation simulation through one week following the end of radiation treatment
  Interventions: Device: wearable sensor
- Primary surgery w/o radiotherapy (Experimental): Patients with head and neck cancer require primary surgery alone (Cohort B-SA)
  A wearable sensor device will be issued at the time of trial enrollment. Patients will be instructed to wear the device on their wrist for 23 hours per day, 7 days per week, from one week before surgery through 1 month following surgery
  Patients with head and neck cancer require primary surgery and postoperative radiotherapy (Cohort B-RT)
  A wearable sensor device will be issued at the time of trial enrollment. Patients will be instructed to wear the device on their wrist for 23 hours per day, 7 days per week, from one week before surgery to one week following the end of radiation treatment .
  Interventions: Device: wearable sensor

INTERVENTIONS:
Device: wearable sensor — A commercially-available wearable fitness sensor
  Other Names: FITBIT

SUMMARY:
The investigator will seek to determine the feasibility of wearable biometric sensors to acquire high resolution biometric data, including heart rate and activity level (i.e. steps) for patients undergoing radiation therapy and surgery, with or without postoperative radiotherapy.

DETAILED DESCRIPTION:
Active cancer treatment such as surgery, chemotherapy or radiotherapy can cause side effects or toxicities, which, if untreated, can lead to poorer quality of life, decreased patient well-being, and worse clinical outcomes. Routine monitoring of patients while under active treatment can entail the routine practice of clinic visits at regular intervals with the acquisition of vital signs, routine laboratory testing, patient-reported outcome surveys, and face-to-face interaction with their physician.

In recent years, the availability of commercially-available wearable fitness sensors has allowed end-users to monitor their fitness progress and activity levels. These devices depend on small sensors that can collect minute-to-minute data on heart rate and activity level that may be transmitted to a smartphone or computer. Through this system, users can easily track and monitor their fitness progress.

In this trial, the investigator will seek to determine the feasibility of wearable biometric sensors to acquire high resolution biometric data, including heart rate and activity level (i.e. steps) for patients undergoing radiation therapy and surgery, with or without postoperative radiotherapy. The investigator believe that changes in heart rate may predict for increasing pain, dehydration, and stress in general. Moreover, changes in daily step count are a surrogate for performance status on treatment, and the investigator will perform a series of preliminary analyses to assess whether there is validity to this hypothesis. The investigator hope to use biometric monitoring to identify patients at risk for adverse outcomes, with the ultimate goal of intervening before these outcomes occur.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven malignancy requiring chemoradiation therapy to the head and neck, OR primary surgery to the head and neck, with or without adjuvant radiotherapy or chemoradiotherapy.
2. Age ≥ 18 years.
3. Performance status ECOG 0-2

   Per typical radiotherapy policy, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry.

   3.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
4. Concurrent chemotherapy is required for definitive radiotherapy patients
5. Hypofractionated or stereotactic body radiation therapy is not permitted
6. Ability to understand and the willingness to sign a written informed consent
7. Willingness to download the Fitbit App to a personal mobile device

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who could wear the device more than 90% of the time, of 23 hours a day, daily | 3 months
  To determine the feasibility of using a commercially-available wearable sensor to obtain biometric data for patients undergoing head and neck locoregional therapy throughout the duration of radiation treatment (cohorts A, B-RT) and throughout post-surgical recovery with or without adjuvant radiotherapy (cohort B)
Daily data acquisition rate | 3 months
  Percentage of successful data acquisition events as well as a retention rate of all enrolled participants.

SECONDARY OUTCOMES:
Changes in daily steps taken | 3 months
  Data will be collected using the Fitbit device and aggregated using the Fitabase platform throughout the duration of radiation treatment (cohorts A, B-RT) and throughout post-surgical recovery with or without adjuvant radiotherapy (cohort B).
Changes in heart rate | 3 months
  Data will be collected using the Fitbit device and aggregated using the Fitabase platform throughout the duration of radiation treatment (cohorts A, B-RT) and throughout post-surgical recovery with or without adjuvant radiotherapy (cohort B).
Changes in sleep habits | 3 months
  Data will be collected using the Fitbit device and aggregated using the Fitabase platform throughout the duration of radiation treatment (cohorts A, B-RT) and throughout post-surgical recovery with or without adjuvant radiotherapy (cohort B).
Volume of intravenous fluids | 3 months
  To analyze associations between biometric parameters and complications and interventions by the volume of intravenous fluids required for patients undergoing radiation treatment (cohorts A, B-RT) and surgical recovery +/-adjuvant radiotherapy (cohort B).
Days of inpatient hospitalization | 3 months
  To analyze associations between biometric parameters and complications and interventions days of inpatient hospitalization required for patients undergoing radiation treatment (cohorts A, B-RT) and surgical recovery +/-adjuvant radiotherapy (cohort B).
Changes in pain level | 3 months
  To analyze associations between biometric parameters and complications and interventions by changes in pain level of patients undergoing radiation treatment (cohorts A, B-RT) and surgical recovery +/-adjuvant radiotherapy (cohort B).
  Pain assessments are based on self-report. Pain scale from 0 no pain, 1-3 minor pain, 4-6 moderate pain to 7-10 severe pain.
Number of emergency department visits. | 3 months
  To analyze associations between biometric parameters and complications and interventions number of emergency department visits required for patients undergoing radiation treatment (cohorts A, B-RT) and surgical recovery +/-adjuvant radiotherapy (cohort B).
Utilization of pain medication | 3 months
  To analyze associations between biometric parameters and complications and interventions utilization of pain medication required for patients undergoing radiation treatment (cohorts A, B-RT) and surgical recovery +/-adjuvant radiotherapy (cohort B).
  Medication Quantification Scale (MQS) Version III will be used to determine drug detriment weight and dosage level.
Physical and mental well-being | 3 months
  To analyze associations between biometric parameters and patient-reported outcomes in regards to physical and mental well-being using the Functional Assessment of Cancer Therapy - General (FACT-G) Health Survey at each weekly scheduled visit to monitor for acute changes in their condition.
Sleep quality | 3 months
  To analyze associations between biometric parameters and patient-reported outcomes in regards to sleep quality using the Pittsburgh Sleep Quality Index (PSQI)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval.

CONTACTS AND LOCATIONS:
Overall Officials: David Sher, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States